CLINICAL TRIAL: NCT02233166
Title: Obstructive Sleep Apnea in Children Referred for Adenotonsillectomy
Brief Title: OSA in Children Referred for Adenotonsillectomy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Lovisenberg Diakonale Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2012/1117
Record Dates: First submitted 2014-08-13; First posted 2014-09-08 (Estimated); Last update posted 2017-08-23 (Actual); Status verified 2015-09

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sample
Oversight: Data Monitoring Committee: No

SUMMARY:
In children with OSA (Obstructive sleep apnea) adenotonsillectomy is regarded as the first choice of treatment. Studies in recent years have shown that the procedure does not always have the expected effect. Children with OSA are at greater risk for complications from the procedure.

There is disagreement regarding the need for sleep studies in children prior to surgery in order to verify an OSA diagnosis. Today less than 10% of these children have polysomnography (PSG).

The main purpose of this study is to describe the prevalence of OSA among children referred for adenotonsillectomy.

The investigators will also examine these children prior to and six months after surgery to assess their sleep pattern and quality of life.

The project outcome aims to improve the precision and quality of diagnosis and the short and long term effects of treatment of children with OSA.

ELIGIBILITY:
Inclusion Criteria:

* age 2-5 year
* referred for adenoidectomy and/or tonsillectomy

Exclusion Criteria:

* craniofacial anomalies
* neurological diseases
* neuropsychiatric diseases

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children aged between 2 and 5 years who are referred for adenoidectomy and/or tonsillectomy.
Sampling Method: Probability Sample
Enrollment: 115 (Estimated)
Dates: Start 2014-08; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Prevalence of OSA | Up to 2 years
  Apne hypopne index (AHI)/ respiratory disturbance index (RDI)

SECONDARY OUTCOMES:
Post operative PSG results | Up to 2 years
  Apne hypopne index (AHI)/ respiratory disturbance index (RDI)

OTHER OUTCOMES:
Quality of life | Up to 2 years
  Questionnaire
Risk factors of OSA | Up to 2 years
  Questionnaire
Post operative complications | Up to 2 years
  Questionnaire; pulse oximetry

CONTACTS AND LOCATIONS:
Locations (1):
- Lovisenberg Diakonale Hospital, Oslo, Norway

REFERENCES:
- [Derived] Overland B, Berdal H, Akre H. Correlations between disease-specific quality of life and polysomnographic findings in children with obstructive sleep apnea. Int J Pediatr Otorhinolaryngol. 2020 Jul;134:110077. doi: 10.1016/j.ijporl.2020.110077. Epub 2020 Apr 30. PMID 32402922